CLINICAL TRIAL: NCT04859985
Title: Selution DeNovo - A Prospective Randomized, Multi-centre, International, Open Label, Clinical Trial Comparing the Selution DEB Strategy Versus DES Strategy.
Brief Title: The SELUTION DeNovo Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.A. Med Alliance S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2021-02
Record Dates: First submitted 2021-03-23; First posted 2021-04-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: Drug Eluting Balloon; Coronary; De Novo coronary lesions
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SELUTION SLR DEB (Experimental): Device: SELUTION SLR DEB. For patients randomized to the DEB strategy, all target lesions should be treated with DEB after appropriate lesion preparation, but provisional DES implantation is acceptable if the angiographic result is considered insufficient either after lesion preparation of after DEB treatment (poor flow, dissection type C or higher, residual stenosis > 30%). For bifurcation lesions, when both main and side- branch are considered to require treatment, a DEB should be used for both.
  Interventions: Device: SELUTION SLR
- DES (Other): Device: Drug Eluting Stent. For patients randomized to the DES strategy, all target lesions should be treated with DES, but use of a SELUTION SLR™ DEB or any other device is acceptable if a DES cannot be delivered to the target lesion. For bifurcation lesions, if the side-branch requires treatment it should be treated with another DES or with POBA, at the discretion of the operator, but not with a DEB.
  Interventions: Device: DES

INTERVENTIONS:
Device: SELUTION SLR — Patients randomized to the SELUTION SLR™ DEB arm will receive lesion preparation according to the 3rd DCB consensus (optimal balloon angioplasty with adjunct treatment using high-pressure balloon, shockwave, rotational atherectomy or cutting or scoring balloon at the discretion of the operator when necessary to maximize lumen diameter). Patients with lesions that are then best treated by provisional stenting (flow-limiting dissection, residual stenosis > 30% or FFR < 0.8) before or after use of DEB will receive a DES but remain in the SELUTION SLR™ DEB group (intention to treat analysis).
  Arms: SELUTION SLR DEB
Device: DES — For patients randomized to the DES strategy, all target lesions should be treated with DES, but use of a SELUTION SLR™ DEB or any other device is acceptable if a DES cannot be delivered to the target lesion. For bifurcation lesions, if the side-branch requires treatment it should be treated with another DES or with POBA, at the discretion of the operator, but not with a DEB.
  Arms: DES

SUMMARY:
A Prospective Randomized, Multi-centre, International, Open Label, Clinical trial comparing the Selution DEB strategy versus DES strategy.

DETAILED DESCRIPTION:
Randomized, multi-centre, international, open label, clinical trial. Patients meeting eligibility criteria will be randomized 1:1 to treatment of all lesions of the identified trial target vessel(s) with either the SELUTION SLR DEB or DES.

Patients randomized to the SELUTION SLR DEB arm will receive lesion preparation according to the 3rd DCB consensus (optimal balloon angioplasty with adjunct treatment using high-pressure balloon, shockwave, rotational atherectomy or cutting or scoring balloon at the discretion of the operator when necessary to maximize lumen diameter). Patients with lesions that are then best treated by provisional stenting (flow-limiting dissection, residual stenosis > 30% or FFR < 0.8) before or after use of DEB will receive a DES but remain in the SELUTION DEB group (intention to treat analysis).

Patients randomized to the DES arm will receive treatment using any CE-marked DES, as per standard institutional practice. Patients with failure to deliver DES will be first treated by provisional DEB using the SELUTION DEB, and failing that, with any other device deemed appropriate.

Staged procedures are allowed if they are planned less than 45 days after the index procedure and are done according to the initial treatment allocation for all trial target vessels (DEB if DEB arm, DES if DES arm).

The study will test:

1. for non-inferiority of a DEB plus provisional DES treatment strategy versus a systematic DES strategy with respect to the primary endpoint of TVF at 12 months.
2. for non-inferiority of a DEB plus provisional DES treatment strategy versus a systematic DES strategy with respect to the primary endpoint of TVF at 5 years. If non-inferiority is then established, superiority of the DEB strategy with TVF as an endpoint will be tested.

All Patients will be followed for clinical outcomes at 30 days, 6 months, 1 2, 3, 4 and 5 years.

ELIGIBILITY:
Subjects must meet all the following criteria to participate in the trial:

* Subject age is ≥ 18 years (or 21 according to countries legal age)
* Female subjects of childbearing potential have a negative pregnancy test ≤7 days before the procedure or are using a contraceptive device or drug.
* Documented angina and/or positive functional testing or unstable angina or stabilized NSTEMI presentation.
* Life expectancy >1 year
* Written informed consent by the subject or her/his legally authorized representative for participation in the study
* One or more native target vessel (LAD, LCX or RCA) is considered to require intervention and is suitable for treatment of all lesions with either DEB + provisional stenting or with DES and is identified as such.
* The number of trial target lesions is not limited, but in the operator's opinion, if the subject is randomized to the DEB arm, the likelihood of the subject requiring provisional stenting of any of the identified trial target lesions is < 30%, and if randomized to the systematic DES arm, all lesions are considered amenable to stenting.
* All target lesions: diameter between 2.0 and 5 mm, and diameter stenosis >50% and <100% with distal flow at least TIMI 2

Exclusion Criteria:

Age < 18 years (or 21 according to countries legal age)

* Subject is pregnant or breast-feeding
* Definite or suspected clinically active covid-19 infection
* Subject is under judicial protection, tutorship or curatorship (for France only)
* Subject is unable to fully comply with the study protocol
* Contraindications to dual antiplatelet therapy, sirolimus or its analogues
* Presentation with STEMI
* Presentation with NSTEMI and ongoing chest pain or hemodynamic instability
* Presentation with Killip III (pulmonary oedema) or IV (cardiogenic shock)
* Chronic NYHA class III or IV heart failure prior to index PCI
* Known LVEF < 30% prior to index PCI
* Previous PCI of a trial target vessel at any time
* Previous PCI of a non-trial target vessel within 30 days
* Trial target lesion located in the left main or any arterial or venous graft
* Trial target lesion is chronic total occlusion (CTO) or in-stent restenosis (ISR)
* Subject considered not able to tolerate at least 30 seconds of coronary occlusion for each trial target lesion
* RVD of trial target lesion > 5mm
* Planned major surgery within one month following the procedure
* Currently participating in another investigational drug or device study that has not completed primary endpoint follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3326 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
TVF | 1 year after treatment
  - TVF (cardiac death, target-vessel related myocardial infarction (MI) or clinically driven target vessel revascularization (cd-TVR) at 1 year
TVF | 5 years after treatment
  - TVF (cardiac death, target-vessel related myocardial infarction (MI) or clinically driven target vessel revascularization (cd-TVR)) at 5 years

SECONDARY OUTCOMES:
Death or any MI | 30 days after treatment
  Cardiac death, non-cardiac death, or any Myocardial Infarction
CD-TVR | 30 days after treatment
  Clinically driven - Target Vessel Revascularization
TVF | 2, 3, 4, 5 years after treatment
  Target Vessel Failure
Any revascularization | 30 days, 6 months, 1, 2, 3, 4 and 5 years after treatment
  1. Target lesion revascularization (TLR) - any and clinically driven
  2. Target vessel revascularization (TVR) - any and clinically driven
  3. A new lesion revascularization in a target vessel
  4. Non-Target vessel revascularization
Myocardial Infarction (MI) | 30 days, 6 months, 1, 2, 3, 4 and 5 years after treatment
  1. Peri-procedural MI
  2. Target-vessel MI
  3. Non-target-vessel MI
  4. MI type (1 to 5) according to the 4th universal definition
Composite of cardiac death or target vessel MI | 30 days, 6 months, 1, 2, 3, 4 and 5 years after treatment
  Composite of cardiac death or target vessel Myocardial Infarction
All-cause mortality | 30 days, 6 months, 1, 2, 3, 4 and 5 years after treatment
  * Cardiac mortality
  * Non-cardiac mortality
Patient-oriented ARC-2 composite endpoint | 30 days, 6 months, 1, 2, 3, 4 and 5 years after treatment
  1. All-cause mortality
  2. Any stroke
  3. Any MI (includes non-target vessel territory)
  4. Any revascularization
Site-reported stroke | 30 days, 6 months, 1, 2, 3, 4 and 5 years after treatment
  Site-reported stroke
Site-reported BARC 3-5 Bleeding | 30 days, 6 months, 1, 2, 3, 4 and 5 years after treatment
  Site-reported BARC (Bleeding Academic Research Consortium ) 3-5 Bleeding
Cost-effectiveness of DEB vs. DES after 12 months in selected countries | 1, 2, 3, 4 and 5 years after treatment
  Total costs of materials used during treatment
Cost-effectiveness of DEB vs. DES after 12 months in selected countries | 1, 2, 3, 4 and 5 years after treatment
  Time of procedure. Total minutes from patient introducer introduction until removal
Cost-effectiveness of DEB vs. DES after 12 months in selected countries | 1, 2, 3, 4 and 5 years after treatment
  Total hospitalization days per procedure.
Net clinical benefit, a combination of freedom from TVF and/or BARC 3-5 bleeding | 30 days, 6 months, 1, 2, 3, 4 and 5 years after treatment
  Net clinical benefit, a combination of freedom from (Target Vessel Failure) TVF and/or BARC 3-5 bleeding
Device success | 30 days, 6 months, 1, 2, 3, 4 and 5 years after treatment
  Device success defined as achievement of a final residual diameter stenosis of < 30% (site-reported), using the assigned device only
Lesion success | 30 days, 6 months, 1, 2, 3, 4 and 5 years after treatment
  Lesion success defined as achievement of < 30% residual stenosis (site-reported), using any PCI method
Procedure success | 30 days, 6 months, 1, 2, 3, 4 and 5 years after treatment
  Procedure success defined as achievement of a final diameter stenosis of < 30% (site-reported) using any PCI method, without the occurrence of death, MI, or repeat target vessel revascularization during hospital stay

CONTACTS AND LOCATIONS:
Locations (62):
- Austria (3):
  - Academic Teaching Hospital Feldkirch, Feldkirch
  - University Heart Center Graz, Graz
  - Kepler Universitätsklinikum GmbH, Linz
- Czechia (2):
  - University Hospital Brno, Brno
  - University Hospital Ostrava, Ostrava
- SIUN sote Hospital and Healthcare center, Joensuu, Finland
- France (6):
  - CH La Rochelle, La Rochelle
  - Hôpital Jaques Cartier, Massy
  - CHU de Nîmes, Nîmes
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier de Pau, Pau
  - Clinique Saint Hilaire, Rouen
- Germany (14):
  - Universitätsklinik Augsburg, Augsburg
  - Universitätsklinikum Freiburg, Bad Krozingen
  - BG Klinikum Unfallkrankenhaus Berlin, Berlin
  - Charite Campus Virchow Klinikum, Berlin
  - Kardiologisch-Angiologische Praxis • Herzzentrum Bremen, Bremen
  - RKH Kliniken Bruchsal Fürst Stirum Klinik, Bruchsal
  - University Koeln, Cologne
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Elisabeth-Krankenhaus, Essen
  - Asklepios Kliniken GmbH & Co., Hamburg
  - University Medical Center Hamburg Eppendorf, Hamburg
  - MEDICLIN Herzzentrum Lahr, Lahr
  - Johannes Wesling Klinikum Minden, Minden
  - Herzklinikum Ulm, Ulm
- Italy (4):
  - Ospedale Civile Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Clinica Mediterranea, Napoli
  - Ospedale Santa Croce di Moncalieri, Torino
  - Ospedale Sant'andrea, Vercelli
- Netherlands (4):
  - University Medical Center Amsterdam, Amsterdam
  - University Medical Center Groningen, Groningen
  - Tergooi MC, Hilversum
  - UMC Utrecht, Utrecht
- Poland (3):
  - Szpital Kliniczny Przemienienia Pańskiego UM, Poznan
  - Kliniczny Szpital Wojewódzki Nr. 2 w Rzeszowie, Rzeszów
  - Szpital Ministerstwa Spraw Wewnetrznych, Rzeszów
- Singapore (2):
  - National Heart Centre Singapore (NHCS), Singapore
  - SengKang General Hospital, Singapore
- Spain (3):
  - Hospital Clinico de Barcelona, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Alvaro Cunqueiro, University Hospital of Vigo, Vigo
- Switzerland (6):
  - University Hospital Basel, Basel
  - University Hospital of Bern, Bern
  - Hôpital Cantonal de Fribourg, Fribourg
  - University Hospital Geneva (HUG), Geneva
  - HOCH Health Ostschweiz Kantonsspital St.Gallen, Sankt Gallen
  - University Zurich, Zurich
- United Kingdom (14):
  - University Hospitals of North Midlands, Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - The Royal Bournemouth and Christchurch Hospitals, Bournemouth
  - Royal Sussex County Hospital, Brighton
  - University Hospitals Bristol, Bristol
  - Royal Infirmary of Edinburgh, Edinburgh
  - Golden Jubilee National Hospital, Glasgow
  - Glenfield Hospital, Leicester
  - Manchester University NHS Foundation Trust, Manchester
  - Norfolk and Norwich University Hospitals, Norwich
  - Trent Cardiac Centre, Nottingham City Hospital, Nottingham
  - Royal Berkshire Hospital, Reading
  - Northern General, Sheffield, Sheffield
  - University Hospital Southampton, Southampton
  - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spaulding C, Krackhardt F, Bogaerts K, Urban P, Meis S, Morice MC, Eccleshall S. Comparing a strategy of sirolimus-eluting balloon treatment to drug-eluting stent implantation in de novo coronary lesions in all-comers: Design and rationale of the SELUTION DeNovo Trial. Am Heart J. 2023 Apr;258:77-84. doi: 10.1016/j.ahj.2023.01.007. Epub 2023 Jan 13. PMID 36642225